CLINICAL TRIAL: NCT01292187
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial Evaluating the Safety and Efficacy of Oral Recombinant Salmon Calcitonin (rsCT) in the Prevention of Postmenopausal Osteoporosis in Women at Increased Risk of Fracture
Brief Title: A Study of Oral Recombinant Salmon Calcitonin (rsCT) to Prevent Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TAR-01-201
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Osteopenia
Keywords: Osteoporosis; Osteopenia; Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Bone Diseases; Musculoskeletal Diseases; Salmon calcitonin; Calcitonin
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral calcitonin at dinner-or bedtime (Experimental): Intervention: Oral calcitonin at dinnertime or oral calcitonin at bedtime. Postmenopausal subjects with osteopenia were treated for one year (also with vitamin D and calcium supplements) to determine if oral calcitonin tablets would prevent the loss of bone mineral density compared with placebo. Randomization to active or placebo was done 2:1. After randomization, further randomization was done to divide each arm into two groups, one in which dosing was at dinnertime and the other in which dosing was at bedtime to determine if food affected efficacy or safety.
  Interventions: Drug: Oral calcitonin at dinnertime; Drug: Oral calcitonin at bedtime
- Oral placebo at dinner- or bedtime (Experimental): Intervention: oral placebo at dinnertime or oral placebo at bedtime
  Interventions: Drug: Oral placebo at dinnertime; Drug: Oral placebo at bedtime

INTERVENTIONS:
Drug: Oral calcitonin at dinnertime — Oral calcitonin at dinnertime.
  Other Names: Oral rsCT
  Arms: Oral calcitonin at dinner-or bedtime
Drug: Oral placebo at dinnertime — Oral placebo at dinnertime.
  Other Names: Placebo
  Arms: Oral placebo at dinner- or bedtime
Drug: Oral calcitonin at bedtime — Oral calcitonin at bedtime
  Other Names: Oral rsCT
  Arms: Oral calcitonin at dinner-or bedtime
Drug: Oral placebo at bedtime — Oral placebo at bedtime
  Other Names: Placebo
  Arms: Oral placebo at dinner- or bedtime

SUMMARY:
The primary purpose of this study was to evaluate the efficacy of oral calcitonin (rsCT)tablets in the prevention of bone loss in postmenopausal women with lower bone mineral density at increased risk of fracture. The secondary purpose of this study was to determine if there is any food effect by comparing the efficacy and safety of oral calcitonin tablets administered at dinner or at bedtime.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled Phase 2 study conducted entirely in the US. The subjects were all post-menopausal women whose 10-year risk of major osteoporotic fracture was assessed using the World Health Organization (WHO) Fracture Risk Assessment Tool (FRAX®) algorithm within the first 3 visits. Eligible, consenting subjects were then enrolled and began a 2- week single-blind placebo run-in phase to determine tolerability. After the run-in phase, continuing subjects were randomized in a 2:1 ratio to receive oral calcitonin or placebo. All subjects took 600 mg calcium citrate and 1000 IU vitamin D once daily with breakfast beginning with the run-in phase. The duration of treatment including the run-in phase was 54 weeks. Bone mineral density (BMD) and C-terminal telopeptide of type 1 collagen (CTx-1) were determined at Baseline and Weeks 28 and 54 after randomization. The % change from baseline in lumbar spine BMD was calculated and compared: active to placebo. The change from baseline in plasma CTx-1 was also calculated and compared likewise.

To confirm that there is no effect of meal timing on this product, subjects in both arms were further randomized to take the active or placebo on an empty stomach at bedtime or with the meal at dinnertime.

ELIGIBILITY:
Inclusion Criteria:

* Female and at least 45 years of age.
* Must have undergone the onset of spontaneous or surgical menopause more than 5 years prior to entry. Spontaneous menopause is defined as 12 months of spontaneous amenorrhea. Surgical menopause is defined as ≥ 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Serum follicle-stimulating hormone (FSH) levels must be ≥ 30 mIU/mL.
* A body mass index (BMI) of not greater than 35 (BMI

  =weight [kg]/height[m]2).
* Bone mineral density (BMD) T-score between -1.0 and - 2.5 at the total hip, femoral neck, trochanter, or lumbar spine.
* Additional risk factors such that the 10 year risk of a major osteoporotic fracture or hip fracture risk is at least as great as a 65-year-old woman of the same race and BMI of 25 kg/m2 as determined by the FRAX algorithm .
* No clinically significant abnormal findings in the medical history or physical exam that would preclude participation in the investigator's opinion.
* No clinically significant abnormal laboratory values at the screening assessment.
* Subjects must give written informed consent after reading the Subject Information and Consent Form and having had the opportunity to discuss the study with the investigator.

Exclusion Criteria:

* History of an osteoporotic fracture, defined as a fracture at the wrist, hip, or humerus occurring from a fall at standing height or less.
* BMD T-Score at any site ≤ -2.5.
* Current treatment (or within 3 months prior to randomization) with hormone replacement therapy.
* History of metabolic and other bone diseases, including osteogenesis imperfecta, osteomalacia, and Paget's disease.
* Vitamin D insufficiency defined as a 25 hydroxyvitamin D level < 20 ng/mL (50 nmol/L).
* Prior use of calcitonin, ever.
* Prior use of any bisphosphonate, ever.
* Prior use of denosumab, fluoride, or strontium, ever.
* Prior use of parathyroid hormone analogs, ever.
* Any condition or disease that may interfere with the ability to have a dual energy x-ray absorptiometry (DXA) scan or to evaluate a DXA scan, for example, severe osteoarthritis of the spine, spinal fusion, pedicle screws, history of vertebroplasty, or degenerative disease that results in insufficient number of evaluable lumbar vertebrae, bilateral hip replacements.
* Use of anabolic steroids or androgens within 6 months preceding randomization.
* Use of vitamin D metabolites and analogs, (e.g., calcitriol) within 3 months preceding randomization). Note: Vitamin D supplementation is not exclusionary.
* Use of estrogen or estrogen-related drugs (including selective estrogen receptor molecules), for example, tamoxifen, tibolone, or raloxifene within 3 months preceding randomization.
* Chronic systemic treatment with glucocorticoids.
* Clinically relevant abnormal history, physical findings, or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the subject.
* Presence of acute or chronic illness or history of chronic illness which, in the judgment of the investigator, makes participation in the study medically inappropriate.
* Known acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV) seropositivity.
* Uncontrolled hypertension, significant gastrointestinal abnormalities, uncontrolled diabetes mellitus, significant coronary heart disease, any psychotic mental illness, chronic allergic rhinitis, asthma, uncorrected endocrine dysfunction, or significantly impaired hepatic, respiratory, or renal function.
* Participation in any other clinical study within the previous month.
* History of drug or alcohol abuse, or intake of more than 30 units of alcohol weekly.
* Possibility that the subject will not cooperate with the requirements of the protocol.
* Known sensitivity to sCT.
* Shift workers-individuals who are at work during overnight hours.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Krause, MD, Study Director — Chief Medical Officer - Tarsa Therapeutics, Inc.
Locations (10):
- United States (10):
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Bethesda Health Research, Bethesda, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Michigan Bone and Mineral Clinic, Detroit, Michigan
  - The Osteoporosis Center at St. Luke's Hospital, Chesterfield, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - University of Pittsburgh - Department of Neurology, Pittsburgh, Pennsylvania
  - Puget Sound Osteoporosis Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- See also: Related Info. — http://www.tarsatherapeutics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from outpatient populations associated with health care centers that treat osteoporosis. Community advertising may also be used for those not associated with such centers.
  Recruitment began on 17 January 2011.
Pre-assignment Details: All patients had a two-week single-blind oral placebo (at bedtime) run-in period before group assignment. This was to accustom the patients to the oral dose regimen prior to randomization
Groups:
- Oral rsCT Tablets: Tablets containing 200 μg of recombinant salmon calcitonin, for oral administration. At group assignment the first 60 patients were told to self-administer the tablets once daily at bedtime (Group 1). The remaining patients were told to self-administer once daily at dinner time (Group 2)to determine if there was any food effect. Randomization was done active:placebo, 2:1.
- Oral Placebo Tablets: Identical appearing placebo tablets, without active ingredient At group assignment the first 60 patients were told to self-administer the tablets once daily at bedtime Group 1). The remaining patients enrolled were told to self-administer once daily at dinner time (Group 2)to determine if there was any food effect. Randomization was done active:placebo, 2:1.
Period: Overall Study
Arm/Group | Oral rsCT Tablets | Oral Placebo Tablets
Started | 86 | 43
Completed | 69 | 30
Not Completed | 17 | 13
Not completed — Adverse Event | 10 | 5
Not completed — Withdrawal by Subject | 6 | 5
Not completed — All other reasons | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Lumbar Spine BMD (Bone Mineral Density) T-scores, plasma CTx-1 (collagen type 1 C telopeptide), , FRAX scores, age, race and body weight were compared between the two treatment arms and were found to have similar means, respectively.
Groups:
- rsCT Tablets: Patients who received oral calcitonin as an active treatment
- Placebo Tablets: Patients who did not receive any active treatment, just placebo
- Total: Total of all reporting groups
Arm/Group | rsCT Tablets | Placebo Tablets | Total
Number analyzed (Participants) | 86 | 43 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 14 | 42
  >=65 years | 58 | 29 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (6.90) | 66.6 (5.16) | 67.2 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 43 | 129
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 81 | 41 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 86 | 43 | 129
T-score [Mean (Standard Deviation); unit: T-score] — The National Osteoporosis Foundation suggested that women with osteopenia (T-score between -1.0 and -2.5 Standard Deviations from the BMD mean value of healthy 30-year old women) and additional risk factors should be treated. For entry into this study, the recommendations of the US Preventative Services Task Force (USPSTF) have been adapted, such that subjects with osteopenia (BMD and a 10-year fracture risk at least that of an average risk 65-year-old woman) were included (World Health Organization's Fracture Risk Assessment Tool (FRAX®) [USPSTF, 2010].
  T-score | -1.15 (0.881) | -1.12 (0.864) | -1.14 (0.872)
FRAX Score [Mean (Standard Deviation); unit: percent probability] — FRAX® is a computer based algorithm (http://www.shef.ac.uk/FRAX) that provides models for the assessment of fracture probability in men and women. The approach uses easily obtained clinical risk factors to estimate 10 year fracture probability for a major fracture due to osteoporosis. Major fracture means a clinically apparent fracture of the hip, spine, humerus (upper arm) or wrist.
  percent probability | 11.87 (5.019) | 11.57 (4.468) | 11.77 (4.827)
LS BMD [Mean (Standard Deviation); unit: grams per square centimeter] — LS BMD was determined at baseline with Dual Energy X-ray Absorptionometry (DEXA) scans and expressed as grams/square centimeter. This was used to calculate T-scores and used as the baseline to assess changes.
  grams per square centimeter | 0.940 (0.106) | 0.929 (0.907) | 0.936 (0.102)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.81 (3.765) | 26.77 (5.983) | 26.13 (25.48)
CTx-1 [Mean (Standard Deviation); unit: ng/L] — C-terminal telopeptide-1
  ng/L | 423.95 (219.419) | 417 (119.882) | 421.74 (193.638)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline to Week 54 of Lumbar Spine Bone Mineral Density of Active Compared to Placebo.
Time Frame: Baseline, Week 54
Population: MITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Oral Calcitonin Tablets: Tablets containing 200 μg of recombinant salmon calcitonin, for oral administration. At group assignment the first 60 patients were told to self-administer the tablets once daily at bedtime (Group 1). The remaining patients were told to self-administer once daily at dinner time (Group 2)to determine if there was any food effect. Randomization was done active:placebo, 2:1.
Arm/Group | Oral Calcitonin Tablets | Oral Placebo Tablets
Number analyzed (Participants) | 74 | 35
percent change | 1.03 [0.46 to 1.59] | -0.12 [-0.94 to 0.71]
Statistical Analysis 1: Comparison: Oral Calcitonin Tablets vs Oral Placebo Tablets; Test type: Superiority or Other; p = 0.0265, Mixed Models Analysis

2. Secondary Outcome: Percentage Change From Baseline to Week 54 of Plasma CTx-1 Following rsCT Compared to Placebo.
Time Frame: Baseline, Week 54
Population: MITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Oral rsCT Tablets | Oral Placebo Tablets
Number analyzed (Participants) | 78 | 36
percent change | -11.83 [-22.43 to -1.43] | 8.37 [-7.11 to 23.85]
Statistical Analysis 1: Comparison: Oral rsCT Tablets vs Oral Placebo Tablets; Test type: Superiority or Other; p = 0.0340, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Oral rsCT Tablets | Oral Placebo Tablets
Serious Adverse Events (participants affected / at risk) | 6/86 | 2/43
Other Adverse Events (participants affected / at risk) | 33/86 | 15/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral rsCT Tablets (N=86) | Oral Placebo Tablets (N=43)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) — Malignant melanoma/ Melanoma On Left Eyelid
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) — Laceration/ Cranial Laceration
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) — Acute Hepatitis
Pericardial effusions (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) — Intermittent Fever
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral rsCT Tablets (N=86) | Oral Placebo Tablets (N=43)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 6 (9)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 7 (8)
Abdominal discomfort (Gastrointestinal disorders) | 9 (11) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No